CLINICAL TRIAL: NCT03588910
Title: Ambulatory Gynecologic Surgery: Finding the Optimal Postoperative Opioid Prescription
Brief Title: Ambulatory Gynecologic Surgery: Finding the Optimal Opioid Prescription
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Kari Plewniak, Director, Pelvic Pain clinic. Associate Fellowship Director. Assistant professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-8755
Record Dates: First submitted 2018-02-16; First posted 2018-07-17 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Surgery
Keywords: ambulatory; narcotics; opioids; postoperative; gynecology; laparoscopy; pain; surgery
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen; Oxycodone

STUDY DESIGN:
Intervention Model Description: Patients are randomized to receive one of two prescription regimens.
Who Masked: Outcomes Assessor
Masking Description: The treating provider and the patient know their prescription. The outcomes assessor will be blinded when administering the postoperative surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Number of oxycodone tablets typically prescribed (Active Comparator): Participants will receive a prescription for 10 tablets of 5 mg oxycodone (1 tablet every 6 hours as needed) as well as 50 tablets of acetaminophen 500mg (1-2 tablets every 6 hours as needed) and 25 tablets ibuprofen 600mg (1tablet every 6 hours as needed).
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen 600 mg; Drug: Oxycodone
- Half the number of oxycodone tablets typically prescribed (Experimental): Participants will receive 5 tablets of 5mg oxycodone as well as 50 tablets of acetaminophen 500mg (1-2 tablets every 6 hours as needed) and 25 tablets ibuprofen 600mg (1tablet every 6 hours as needed).
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen 600 mg; Drug: Oxycodone

INTERVENTIONS:
Drug: Acetaminophen — 50 tablets of acetaminophen 500mg (1-2 tablets every 6 hours as needed)
  Other Names: Tylenol
Drug: Ibuprofen 600 mg — 25 tablets ibuprofen 600mg (1tablet every 6 hours as needed)
  Other Names: Motrin
Drug: Oxycodone — The number of tablets of oxycodone prescribed is the only difference between the two arms.

SUMMARY:
Currently there is a nationwide epidemic in opioid abuse and overdose deaths. While the opioid epidemic is multi-factorial one major source of excess opioids may be over-prescribing in the post-operative period. There is wide variation in the prescribing practices for post-operative pain control and there is no standard of care for pain control after minor laparoscopic surgery in general or after gynecologic laparoscopy. There is also evidence to show that on average half of the opioids prescribed are unused by the patient. The aim of the study is to evaluate two opioid prescription regimens.

DETAILED DESCRIPTION:
This will be a randomized controlled study enrolling participants scheduled for outpatient minor laparoscopic gynecologic surgery. This is a two arm study consisting of 60 subjects in each arm. The participants will be randomized at the time of enrollment. We will use computer generated blocks of four participants. Both arms of participants will receive the same non-narcotic pain medication prescriptions which will include fifty tablets of acetaminophen 500mg (1-2 tablets every 6 hours as needed) and twenty-five tablets ibuprofen 600mg (1 tablet every 6 hours as needed). The arms will only differ in the number of tablets of oxycodone prescribed. In one arm (experimental) subjects will receive five tablets of oxycodone 5mg (1 tablet every 6 hours as needed) and the other arm (comparator) ten tablets of oxycodone 5mg (1 tablet every 6 hours as needed). Both prescription regimens are within the range of normal clinical practice for post-operative pain control.

The participants will receive a telephone call by administrative staff, who is not directly involved in the participants care or data collection for the study subjects, on postoperative day 1 and 7. The participants will all be scheduled for a 2- week post-operative follow up with the surgeon in the office. The primary outcome to be assessed will be number of opioids used by the participants at 24 hours and 7 days post-operative. The primary hypothesis is that participants prescribed only 5 tabs of oxycodone will not require more medication. The secondary hypothesis is that the pain scores between the two groups will not be different. The other variables being studied include the following: having had a post-operative bowel movement, presence of nausea, number of ibuprofen, acetaminophen tablets remaining, calls to the office prior to the follow up visit for pain issues, and urgent or emergency department visits for pain issues. These assessments will be asked during the brief telephone calls and also at the postoperative visit.

All participants will be given the clinic phone number and advised to call with any questions or clinical concerns. The participants will be advised if possible to return to a Montefiore Emergency Department or gynecologic provider in case of an urgent issue prior to the 2 week postoperative visit, as opposed to an outside facility.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age
* Scheduled for outpatient gynecologic laparoscopy

Exclusion Criteria:

* Significant renal or liver disease is present that would alter prescribing patterns
* Chronic opioid use or abuse
* Allergy to acetaminophen, ibuprofen, other nsaids or narcotic medications
* Conversion of surgery to exploratory laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ja Hyun Shin, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomazeau J, Rouquette A, Martinez V, Rabuel C, Prince N, Laplanche JL, Nizard R, Bergmann JF, Perrot S, Lloret-Linares C. Acute pain Factors predictive of post-operative pain and opioid requirement in multimodal analgesia following knee replacement. Eur J Pain. 2016 May;20(5):822-32. doi: 10.1002/ejp.808. Epub 2015 Oct 30. PMID 26517014
- [Background] De Oliveira GS Jr, Ahmad S, Fitzgerald PC, Marcus RJ, Altman CS, Panjwani AS, McCarthy RJ. Dose ranging study on the effect of preoperative dexamethasone on postoperative quality of recovery and opioid consumption after ambulatory gynaecological surgery. Br J Anaesth. 2011 Sep;107(3):362-71. doi: 10.1093/bja/aer156. Epub 2011 Jun 13. PMID 21669954
- [Background] As-Sanie S, Till SR, Mowers EL, Lim CS, Skinner BD, Fritsch L, Tsodikov A, Dalton VK, Clauw DJ, Brummett CM. Opioid Prescribing Patterns, Patient Use, and Postoperative Pain After Hysterectomy for Benign Indications. Obstet Gynecol. 2017 Dec;130(6):1261-1268. doi: 10.1097/AOG.0000000000002344. PMID 29112660
- [Background] Baruch AD, Morgan DM, Dalton VK, Swenson C. Opioid Prescribing Patterns by Obstetrics and Gynecology Residents in the United States. Subst Use Misuse. 2018 Jan 2;53(1):70-76. doi: 10.1080/10826084.2017.1323928. Epub 2017 Sep 1. PMID 28862884
- [Background] Darnall B, Li H. Hysterectomy and predictors for opioid prescription in a chronic pain clinic sample. Pain Med. 2011 Feb;12(2):196-203. doi: 10.1111/j.1526-4637.2010.01038.x. Epub 2011 Jan 11. PMID 21223499
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
Started | 60 | 60
Post Op Day 1 Survey | 52 | 47
Completed (Post Op Day 7 Survey) | 47 | 45
Not Completed | 13 | 15
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Allergy | 2 | 0
Not completed — Protocol Violation | 0 | 3
Not completed — Did not complete Day 1 Survey | 5 | 10
Not completed — Did not complete Day 7 Survey | 5 | 2

BASELINE CHARACTERISTICS:
Population: Patients were excluded who withdrew consent, failed the protocol (did not undergo the planned surgery).
Groups:
- Total: Total of all reporting groups
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 57 | 114
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.0) | 37.0 (7.7) | 36.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 32 | 39 | 71
  Non-Hispanic Black | 12 | 9 | 21
  White | 5 | 1 | 6
  Unknown | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Oxycodone Tablets Used Day 1
Description: During the survey phone call on day 1, participants will be asked to report the total number of oxycodone tablets use since the surgery.
Time Frame: 24 hours post-operative
Population: Participants answering Day 1 Survey
Measure: Median (Inter-Quartile Range); unit: Oxycodone Tablets
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
Number analyzed (Participants) | 52 | 47
Oxycodone Tablets | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Number of Oxycodone Tablets Typically Prescribed vs Half the Number of Oxycodone Tablets Typically Prescribed; Test type: Superiority — Wilcoxon rank-sum tests; p = .87, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Oxycodone Tablets Used as Reported by Participants 1 Week After Surgery
Description: During the survey phone call on day 7, participants will be asked to report the total number of oxycodone tablets used since the surgery.
Time Frame: 7 days post-operative
Population: Participants who answered survey on Day 7. Not all participants answered each question on follow up surveys.
Measure: Median (Inter-Quartile Range); unit: Oxycodone Tablets
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
Number analyzed (Participants) | 46 | 44
Oxycodone Tablets | 2.5 [0.0 to 5.0] | 2.0 [0.0 to 4.0]
Statistical Analysis 1: Comparison: Number of Oxycodone Tablets Typically Prescribed vs Half the Number of Oxycodone Tablets Typically Prescribed; Test type: Superiority — Wilcoxon rank-sum tests; p = .36, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Self Reported Pain Score on Post Operative Day 1 (Numeric Pain Reporting Score: NRS)
Description: Participants will be surveyed during the phone call survey to rate pain score on a scale from 0 (no pain), to 10 (severe pain)
Time Frame: 1 day post operative
Population: Participants completing Day 1 Survey
Measure: Median (Inter-Quartile Range); unit: Score on Numeric Pain Scale
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
Number analyzed (Participants) | 52 | 47
Score on Numeric Pain Scale | 5.0 [3.0 to 7.0] | 5 [2.0 to 6.0]
Statistical Analysis 1: Comparison: Number of Oxycodone Tablets Typically Prescribed vs Half the Number of Oxycodone Tablets Typically Prescribed; Test type: Superiority; p = .91, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Self Reported Pain Score on Post Operative Day 7 (Numeric Pain Reporting Score: NRS)
Description: as for outcome 3
Time Frame: 7 days post operative
Population: Participants completing Day 7 Survey
Measure: Median (Inter-Quartile Range); unit: Score on Numeric Pain Scale
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
Number analyzed (Participants) | 47 | 45
Score on Numeric Pain Scale | 2.0 [0.0 to 4.0] | 1.3 [0.0 to 3.3]
Statistical Analysis 1: Comparison: Number of Oxycodone Tablets Typically Prescribed vs Half the Number of Oxycodone Tablets Typically Prescribed; Test type: Superiority; p = .29, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Additional Contacts With Provider
Description: By chart review, unscheduled interactions with the healthcare system related to pain will be counted.These will include phone calls related to pain, unscheduled visits to the office or emergency department
Time Frame: 1 week post operative
Measure: Number; unit: Unscheduled patient contacts
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
Number analyzed (Participants) | 57 | 57
Unscheduled patient contacts | 1 | 4
Statistical Analysis 1: Comparison: Number of Oxycodone Tablets Typically Prescribed vs Half the Number of Oxycodone Tablets Typically Prescribed; Test type: Superiority; p = .36, Chi-squared

ADVERSE EVENTS:
Time Frame: The follow up time included 6 weeks post operative
Description: We used the same definitions.
Arm/Group | Number of Oxycodone Tablets Typically Prescribed | Half the Number of Oxycodone Tablets Typically Prescribed
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03588910/Prot_SAP_000.pdf